CLINICAL TRIAL: NCT01615523
Title: Executive Function in Preterm Born Children: An Integrative Approach From Genetics to Brain Function
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: EF_MRI_EEG
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Preterm Infants
Keywords: Executive functions
MeSH Terms: interventions — Magnetic Resonance Spectroscopy; Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Children/adolescents born preterm
  Interventions: Other: MRI, EEG and cognitive testing
- Control children and adolescents
  Interventions: Other: MRI, EEG and cognitive testing

INTERVENTIONS:
Other: MRI, EEG and cognitive testing — Sleep EEG and one MRI, executive function testing using Strrop test, BRIEF questionnaire and CantabEclipse

SUMMARY:
Hd-EEG and MRI measures are used to study the maturation of functional networks in order to identify the neural circuits underlying executive and memory processes in children born preterm. It will be determined whether children born preterm with executive function deficits will have an abnormal connectivity between basal ganglia and cortex due to WM injury. Moreover, the development of hd-EEG activity during sleep (coherence and travelling waves) and brain maturation of children and adolescents born preterm will be compared with the respective measures in healthy controls. This is of eminent importance as it helps to understand the nature of executive function and hence, it may help to develop neuroprotective strategies to prevent executive function deficits in these infants.

ELIGIBILITY:
Inclusion criteria:

* Schoolchildren between 10 and 12 or 14 and 16 (born between 1996 and 1998 or between 2000 and 2002)
* Preterm group: born <32 weeks of gestation
* Control group: siblings or friends of preterm group in one of the two age groups

Exclusion criteria:

* Preterm Group: MDI < 85 at 5 years of age; cerebral palsy
* Control Group: born <37 weeks of gestation

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children and adolescents born preterm with their peers as controls
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2012-09; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia F Hagmann, MD, Principal Investigator — University Hospital Zurich, Division of Neonatology
Locations (1):
- University Hospital Zurich, Division of Neonatology, Zurich, Canton of Zurich, Switzerland